CLINICAL TRIAL: NCT05433233
Title: Effects of Lifestyle Walking on Blood Pressure in Older Adults With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Duck-chul Lee, Professor, Iowa State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-375-00
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Hypertension; Aging
MeSH Terms: conditions — Hypertension | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAPA (Experimental): Participants assigned additional 3,000 steps/day on 5 days/week. Participants also received an additional 15 minutes of structured conversation with research personnel following the Health Action Process Approach Theory for behavior change.
  Interventions: Behavioral: Walking; Other: HAPA Behavior Change Counseling
- No HAPA (Experimental): Participants assigned additional 3,000 steps/day on 5 days/week and general conversation with researchers in regard to behavior change, not following a structured dialogue.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Walking — Participants will perform 3,000 additional steps/day on 5 days/week.
Other: HAPA Behavior Change Counseling — Structured dialogue for initiating behavior change.
  Arms: HAPA

SUMMARY:
Eight out of ten older adults have hypertension in the US, which is a strong risk factor for cardiovascular events. To manage hypertension, regular and structured exercise is effective and strongly recommended regardless of drug therapy. However, structured exercise is often performed in a health club, could be difficult, and warrants caution in older adults with chronic conditions. In contrast, the most common lifestyle physical activity in older adults is walking, which is inexpensive, easy, and safe. Recent technological advancement in activity monitoring provides reliable step counts and promotes lifestyle walking. Although one of the most popular public health goals is walking 10,000 steps/day, recent studies found that it is unrealistic and difficult to achieve. Further, there is very little evidence whether walking 10,000 steps/day is effective, specifically in older adults with hypertension. Walking 3,000 extra steps/day 5 days/week is equivalent to meeting the current aerobic physical activity guidelines, as it takes about 30 minutes each day, and is more realistic and achievable. Steps/day is easy to understand and captures most physical activities in older adults. However, there are no specific guidelines about how many daily steps are needed for older adults in the current physical activity guidelines. Thus, this project is aimed to provide pilot data to answer a simple, but unknown, question about physical activity in older adults: "Can increasing lifestyle walking in older adults with hypertension reduce blood pressure? And can older adults maintain a lifestyle walking intervention on their own?". This project will significantly contribute to developing more effective and easy physical activity guidelines for older adults.

DETAILED DESCRIPTION:
All participants will be prescribed a step goal to increase their walking by 3,000 steps/day on 5 days/week for 20 weeks. During the first 10 weeks, support will be provided by research personnel to actively help obtain these goals. During weeks 11-20, participants will be in a self-maintenance phase where no research personnel assistance will be provided to help maintain the extra walking. Participants will log their steps every day during the 20-weeks from a pedometer that they will wear daily. Participants will assess blood pressure and weight at baseline, 10 and 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 65+
* Systolic/diastolic blood pressure of 130-159/80-99 mmHg. Participants will be allowed to be on blood pressure medication.
* Body mass index of 25-40 kg/m2
* Non-smokers
* Sedentary/inactive individuals: not meeting the current aerobic physical activity guidelines of 150 minutes per week over the past 3 months
* Baseline average daily step count <8,000 steps

Exclusion Criteria:

* Any significant mobility limitation because our intervention requires an increase in 3,000 steps per day, which needs to be achievable by the participant.
* A stroke, myocardial infarction (heart attack) or cancer diagnosis within the last 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | 20 weeks
  The primary outcome is the change in measured systolic and diastolic blood pressure from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Duck-chul Lee, PhD, Principal Investigator — Iowa State University
Locations (1):
- Iowa State University, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Request for sharing de-identified data should be addressed to the Principal Investigator: Duck-chul Lee at dclee@iastate.edu
Supporting Information: SAP, ICF
Time Frame: One year after publication
Access Criteria: With a signed data use agreement with Iowa State University